CLINICAL TRIAL: NCT05541887
Title: Acute and Chronic Impacts of Muscadine Wine Polyphenols on Cognition, Memory, Mood, and Anxiety in Adults Over 50 Years of Age
Brief Title: Use Muscadine Wine Nutraceuticals to Improve Brain Health, Cognition, and Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB202300014
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Performance; Memory; Mood; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Placebo (Active Comparator): Participants in this arm will consume muscadine wine polyphenol for six weeks and then placebo for another six weeks. The two phases are separated by a 21-day washout period
  Interventions: Other: Muscadine Wine Polyphenol; Other: Placebo
- Placebo-Intervention (Active Comparator): Participants in this arm will first consume placebo for six weeks and then muscadine wine polyphenol for another six weeks. The two phases are separated by a 21-day washout period
  Interventions: Other: Muscadine Wine Polyphenol; Other: Placebo

INTERVENTIONS:
Other: Muscadine Wine Polyphenol — dealcoholized muscadine wine with alcohol content <0.5% with addition of 50ppm of sodium metabisulfite for preservation
  Other Names: Dealcoholized Muscadine Wine
Other: Placebo — this placebo beverage is formulated with matching sugar and organic acid content to the muscadine wine polyphenol. Food coloring is added to match the color of the intervention. 50ppm of sodium metabisulfite for preservation

SUMMARY:
Previous studies have shown that polyphenol-rich foods can positively affect cognitive functions, memory, and mood in humans. We hypothesize that both acute and chronic intake of muscadine wine polyphenols will improve cognitive performance and mood through regulating the HPA axis, alleviating inflammation and oxidative stress, and/or inhibiting monoamine oxidase activities

DETAILED DESCRIPTION:
Although the exact biological mechanisms for depression and Alzheimer's Disease are not fully understood, it's believed that they are caused by a combination of factors. An increasing amount of scientific research has proposed several possible pathophysiologies linking depression and AD. For example, increased production of pro-inflammatory cytokines in the nervous system, oxidative stress induced by chronic inflammation leads to dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis, and disturbance in the brain-derived neurotrophic factor signal pathway. Polyphenol has been well recognized for its antioxidant and anti-inflammatory properties. Previous studies have shown that polyphenol-rich food such as concord grape juice, blueberries, blackcurrants, and green oats positively affect cognition, memory, and mood in humans. However, no one has examined the effects of muscadine wine polyphenol on cognitive and mental health. In addition, if they do have effects, through what mechanism? This clinical trial will allow us to investigate the questions raised. We hypothesize that intake of muscadine wine polyphenols enhances cognition and memory and improve depression and anxiety in healthy adults over 50 year-old via regulating the HPA axis, alleviating inflammation and oxidative stress, and/or inhibiting monoamine oxidase activities. The research will provide the first clinical evidence of how muscadine wine polyphenols affect the brain and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI (18.5-29.9)
* Body weight ≥110 pounds

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Smokers
* Diabetic
* Heavy drinkers
* Subjective but not clinically diagnosed cognitive impairment (Montreal cognitive assessment score <26),
* Inability to understand the cognitive function tasks
* Intake of medication that might influence the outcome of the study (e.g. psychostimulant)
* cannabis product user
* Clinically diagnosed mental illnesses
* Cardiovascular and neurological disorders
* Uncontrolled hypertension

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline cognitive performance score after intervention/placebo | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Participants will complete the NIH Toolbox cognitive battery. The test battery incorporates multiple tests that assess various aspects of cognitive performance. The list of tests and the function they measure are the following.1. Flanker inhibitory control and attention test (executive function): scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these vectors ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value 0-10. The higher the score the better the performance. 2. Dimensional Change Card Sort (cognitive flexibility): scoring is the same as Flanker's test.
Change from baseline cognitive performance score after intervention/placebo - continued | Baseline, acute (4-hour post single dose), chronic (end of six week)
  3. Picture Sequence Test (episodic memory): Item Response Theory (IRT) is used to score this test. score known as a theta score is calculated for each participant; it represents the relative overall ability or performance of the participant. A theta score is very similar to a z-score, which is a statistic with a mean of zero and a standard deviation of one. The higher the score, the better the performance. 4. List Sorting Test (working memory: scored by summing the total number of items correctly recalled and sequenced on the tests, which can range from 0-26. 5. Pattern and Comparison Test (processing speed): The participant's raw score is the number of items answered correctly in 85 seconds of response time, with a range of 0-130. higher score means better performance. Both individual test scores and composite scores will be compared to baseline score
Change from baseline cognitive performance score after intervention/placebo - continued | Baseline, acute (4-hour post single dose), chronic (end of six week)
  6. Rey's Auditory Verbal Learning Test assesses immediate and delayed (30min) recall of a given list of words that is repeated 5 times. The number of correct words recalled and intrusion words (extraneous word offered by the participant that does not appear on the list) are recorded for scoring
Change from baseline monoamine oxidase (MAOs) activity | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Blood samples will be drawn immediately after the completion test battery. Blood plasma level of monoamine oxidase (MAOs) activity will be determined using the Amplex Red Monoamine Oxidase Assay Kit to assess the inhibitory effects of muscadine wine/juice on MAOs.
Change from baseline neurotransmitters | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Plasma levels of acetylcholine, dopamine, melatonin, serotonin, epinephrine, and γ-aminobutyric acid (GABA) will be quantified using the targeted metabolomic method on UHPLC-MS/MS
Change from baseline brain-derived neurotrophic factors | Baseline, acute (4-hour post single dose), chronic (end of six week)
  plasma BDNF will be measured using ELISA
Change from baseline cortisol, TNF-α, high sensitivity C-reactive protein, and LPS binding protein | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Plasma levels will be measured using ELISA

SECONDARY OUTCOMES:
Change from baseline mood and anxiety score after intervention/placebo | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Participants will complete the NIH Toolbox emotion battery. The test battery include two self-report measure,
  1. Positive affect survey (assess mood): 5-point scale with options ranging from "not at all" to "very much." higher scores are indicative of more positive affect
  2. Fear-Affect Survey (assess anxiety): 5-point scale with options ranging from "never" to "always." higher scores are indicative of more feelings of fear and anxiety
Change from baseline depression score after intervention/placebo | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Depression score will be assessed with Beck's Depression inventory. The questionnaire consists of 21 items with a four point scale ranges between 0-3. The higher the total score the more severe the depression.
Change from baseline pro-inflammatory cytokines | Baseline, acute (4-hour post single dose), chronic (end of six week)
  Inflammatory response will be evaluated by measuring the plasma level of pro-inflammatory cytokines IL-1beta, IL-6, and TNF-alpha using Elisa Kits

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and human nutrition department at University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menard C, Pfau ML, Hodes GE, Kana V, Wang VX, Bouchard S, Takahashi A, Flanigan ME, Aleyasin H, LeClair KB, Janssen WG, Labonte B, Parise EM, Lorsch ZS, Golden SA, Heshmati M, Tamminga C, Turecki G, Campbell M, Fayad ZA, Tang CY, Merad M, Russo SJ. Social stress induces neurovascular pathology promoting depression. Nat Neurosci. 2017 Dec;20(12):1752-1760. doi: 10.1038/s41593-017-0010-3. Epub 2017 Nov 13. PMID 29184215
- [Background] Du X, Pang TY. Is Dysregulation of the HPA-Axis a Core Pathophysiology Mediating Co-Morbid Depression in Neurodegenerative Diseases? Front Psychiatry. 2015 Mar 9;6:32. doi: 10.3389/fpsyt.2015.00032. eCollection 2015. PMID 25806005
- [Background] Haskell-Ramsay CF, Stuart RC, Okello EJ, Watson AW. Cognitive and mood improvements following acute supplementation with purple grape juice in healthy young adults. Eur J Nutr. 2017 Dec;56(8):2621-2631. doi: 10.1007/s00394-017-1454-7. Epub 2017 Apr 20. PMID 28429081
- [Background] Lamport DJ, Lawton CL, Merat N, Jamson H, Myrissa K, Hofman D, Chadwick HK, Quadt F, Wightman JD, Dye L. Concord grape juice, cognitive function, and driving performance: a 12-wk, placebo-controlled, randomized crossover trial in mothers of preteen children. Am J Clin Nutr. 2016 Mar;103(3):775-83. doi: 10.3945/ajcn.115.114553. Epub 2016 Feb 10. PMID 26864371
- [Background] Whyte AR, Schafer G, Williams CM. Cognitive effects following acute wild blueberry supplementation in 7- to 10-year-old children. Eur J Nutr. 2016 Sep;55(6):2151-62. doi: 10.1007/s00394-015-1029-4. Epub 2015 Oct 5. PMID 26437830
- [Background] Watson AW, Haskell-Ramsay CF, Kennedy DO, Cooney JM, Trower T, Scheepens A. Acute supplementation with blackcurrant extracts modulates cognitive functioning and inhibits monoamine oxidase-B in healthy young adults. Journal of Functional Food. 2015 Aug;17:524-539. doi:10.1016/j.jff.2015.06.005
- [Background] Kennedy DO, Bonnlander B, Lang SC, Pischel I, Forster J, Khan J, Jackson PA, Wightman EL. Acute and Chronic Effects of Green Oat (Avena sativa) Extract on Cognitive Function and Mood during a Laboratory Stressor in Healthy Adults: A Randomised, Double-Blind, Placebo-Controlled Study in Healthy Humans. Nutrients. 2020 May 29;12(6):1598. doi: 10.3390/nu12061598. PMID 32485993
- [Background] Bandaruk Y, Mukai R, Kawamura T, Nemoto H, Terao J. Evaluation of the inhibitory effects of quercetin-related flavonoids and tea catechins on the monoamine oxidase-A reaction in mouse brain mitochondria. J Agric Food Chem. 2012 Oct 17;60(41):10270-7. doi: 10.1021/jf303055b. Epub 2012 Oct 8. PMID 23009399
- [Background] Zhu WL, Shi HS, Wei YM, Wang SJ, Sun CY, Ding ZB, Lu L. Green tea polyphenols produce antidepressant-like effects in adult mice. Pharmacol Res. 2012 Jan;65(1):74-80. doi: 10.1016/j.phrs.2011.09.007. Epub 2011 Sep 22. PMID 21964320
- [Background] Olasehinde TA, Oyeleye SI, Ibeji CU, Oboh G. Beetroot supplemented diet exhibit anti-amnesic effect via modulation of cholinesterases, purinergic enzymes, monoamine oxidase and attenuation of redox imbalance in the brain of scopolamine treated male rats. Nutr Neurosci. 2022 May;25(5):1011-1025. doi: 10.1080/1028415X.2020.1831260. Epub 2020 Oct 15. PMID 33054666